CLINICAL TRIAL: NCT01973478
Title: Deep Brain Stimulation in Patients With Chronic Treatment Resistant Depression
Acronym: STHYM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 35RC08_8902
Record Dates: First submitted 2013-10-08; First posted 2013-10-31 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Major Depressive Disorder; Recurrent Depressive Disorder; Bipolar Disorder
Keywords: Major depressive disorder; Recurrent depressive disorder; Bipolar disorder; Deep brain stimulation; Accumbens
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBS (Experimental): The medical device includes:
  * Either a pacemaker ACTIVA PC (Ref 37601) two-channel (Medtronic USA) or two pacemakers Activa SC (Ref 37603) to a channel (Medtronic USA)
  * Two DBS electrodes with four contacts (type Medtronic DBS 3389). Patients will be operated with the usual stereotactic surgical procedure.
  The target is the Accumbens nucleus.
  The two electrodes are implanted in a single session under local anaesthesia or intermittent sedation (propofol parenteral without intubation early intervention). Day 0 is defined by the surgery.
  The DBS is "on" during 6 months (between Month 1 and Month 7). Stimulation will also be on after Month 7.
  Interventions: Device: DBS
- SHAM (Sham Comparator): The medical device includes:
  * Either a pacemaker ACTIVA PC (Ref 37601) two-channel (Medtronic USA) or two pacemakers Activa SC (Ref 37603) to a channel (Medtronic USA)
  * Two DBS electrodes with four contacts (type Medtronic DBS 3389). Patients will be operated with the usual stereotactic surgical procedure.
  The target is the Accumbens nucleus.
  The two electrodes are implanted in a single session under local anaesthesia or intermittent sedation (propofol parenteral without intubation early intervention). Day 0 is defined by the surgery.
  The DBS is "off" during 6 months (between Month 1 and Month 7). Possibility to active the stimulation after Month 7.
  Interventions: Device: SHAM

INTERVENTIONS:
Device: DBS
  Arms: DBS
Device: SHAM
  Arms: SHAM

SUMMARY:
Major depressive disorders are real public health issues in terms of diagnosis and treatment. Some forms of depression are chronic and resistant to treatment (TRD). In these forms suicide risk is important.

Patients with TRD are potential candidates for neurosurgical interventions to treat depression. However, psychosurgery interventions based upon lesions, showed their limitations related to 1. the large variability in neurosurgical gestures, 2. their side effects, and of course 3. the irreversible damage caused by the surgery.

Thus, deep brain stimulation (DBS) could represent an opportunity for patients suffering from TRD. Our preliminary study based upon the stimulation of the accumbens nucleus showed encouraging results. The investigators have thus planned a randomized controlled trial versus sham stimulation to confirm the therapeutic value of nucleus accumbens DBS.

DETAILED DESCRIPTION:
Because of their recurrent nature, their prevalence and their consequences, major depressive disorders are real public health issues in terms of diagnosis and treatment.

Some forms of depression are chronic and resistant to treatment (TRD), either unipolar (repeated episodes of depression) or bipolar (repeated episodes of depression and manic and/or hypomanic episodes). In these forms suicide risk is important.

Patients with TRD are potential candidates for neurosurgical interventions to treat depression. The benefit of neurosurgical procedures is expected to be important in these patients.

Psychosurgery interventions based upon lesions, however, showed their limitations related to 1/ the large variability in neurosurgical gestures, 2/ their side effects, and of course 3/ the irreversible damage caused by the surgery.

Current brain imaging data yielded fresh information about the pathophysiology of depression and suggested new therapeutic approaches in TRD.

Modulation of sub-caudate specific pathways, which are part of orbitofrontal and anterior cingulate cortico-subcortical loops should allow for a diminution of depressive symptoms.

The modulation of these specific pathways, initially targeted by classical neurosurgery, could benefit from current developments in functional neurosurgery.

Deep brain stimulation (DBS) may represent an opportunity for patients suffering from TRD. Our preliminary study based upon the stimulation of the accumbens nucleus showed encouraging results. The investigators have thus planned a randomized controlled trial versus sham stimulation to confirm the therapeutic value of nucleus accumbens DBS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* DSM-IV (DSM = Diagnostic and Statistical Manual) criteria for a recurrent depressive disorder or bipolar disorder
* Duration of the episode > 2 years
* Severity of the episode attested by :

  * A HDRS score > 21
  * A CGI score ≥ 4
  * A GAF < 50
* Persistence of severity criteria during the screening
* Following characteristics resistance in case of recurrent depressive disorder :

  * Stage V of the classification of Thase and Rush
  * Unsuccessful treatment by the association of two antidepressants (or intolerance/contra-indications)
  * Unsuccessful treatment by the association for at least 6 weeks of one of the following treatments : lithium , thyroid hormone , buspirone , pindolol with an antidepressant (or intolerance/contra-indications)
  * Unsuccessful treatment by the combination of a second-generation antipsychotic (olanzapine, risperidone, amisulpride, aripiprazole, clozapine and quetiapine) to an antidepressant (or intolerance/contra-indications)
  * Unsuccessful treatment by a structured psychotherapy
* Following characteristics of resistance in case of bipolar disorder:

  * Unsuccessful treatment by lithium (or intolerance/contra-indications)
  * Unsuccessful treatment by at least one mood stabilizer anticonvulsant (or intolerance/contra-indications)
  * Unsuccessful treatment by at least one second-generation antipsychotic (or intolerance/contra-indications)
  * Unsuccessful treatment by the combination of two mood stabilizers with at least an anticonvulsant (or intolerance/contra-indications)
  * Unsuccessful treatment by electro-convulsive therapy sessions (or intolerance/contra-indications)
  * Unsuccessful treatment by at least one antidepressant , mood stabilizer combination (or intolerance/contra-indications)
  * Unsuccessful treatment by a structured psychotherapy
* Understanding the conduct of the study
* Giving a written informed consent
* Benefiting from the french social insurance

Non-Inclusion Criteria:

* Comorbid axis 1 disorder (except dysthymia, generalized anxiety disorder, social phobia, panic disorder)
* Alcohol or other psychoactive substances dependence (except nicotine)
* Suicidal risk during the last month assessed by the MINI (Mini International Neuropsychiatric Interview), the DIGS (Diagnostic Interview for Genetic Studies) and the item 3 of the HDRS
* Suicide attempt in the last 6 months or two suicide attempts in the previous two years
* History of forensic act or furious mania
* Depressive episode with congruent or incongruent psychotic features or history of a depressive episode with psychotic features
* Comorbid cluster A or B personality disorders according to the DSM IV-TR evaluated using the SCID2 (Structured Clinical Interview for DSM-IV)
* Cognitive Impairment (Mattis < 130)
* MRI (Magnetic Resonance Imaging) contraindication to stimulation or contraindications for MRI
* Major somatic disease making it impossible to set up the study treatment
* Pregnant women, or nursing or childbearing potential without effective contraception
* Involuntary commitment
* Guardianship
* Participation in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Response = 50 % decrease of the HDRS-17 (Hamilton depression rating scale, 17 items version) (yes/no) | Month 7
  Response is defined as a 50 % decrease of the HDRS-17 (Hamilton depression rating scale, 17 items version)

SECONDARY OUTCOMES:
Remission (yes/no) | Month 7
  Remission is defined as an HDRS-17 score < 7
CGI (Clinical global impressions) amelioration (yes/no) | Month 7
  Score of 1 or 2 (item 2 of the CGI)
GAF (Global assessment of functioning) | Month 7
  Presence of a score ≥ 60
HDRS-17 (Hamilton depression rating scale, 17 items version) | Month 7
  Score
MADRS (Montgomery-Asberg Depression Rating Scale) | Month 7
  Score
BDI (Beck Depression Inventory) | Month 7
  Score
CGI (Clinical global impressions) | Month 7
  Score
LARS (Lille Apathy Rating scale) | Month 7
  Score
GAF (Global assessment of functioning) | Month 7
  Score
Neuropsychological assessment | Day -7 ; Month 1; Month 7; Month 13; Month 19; Month 24
Cerebral metabolism (PET scans) | Day -7; Month 7
Adverse events | Month 24
  Adverse events occuring during the study.

OTHER OUTCOMES:
HDRS-17 (Hamilton depression rating scale, 17 items version) | Month -3 ; Month -1; Day -7; Day 15; Month 1; Day 45; Month 2 ; Day 75 ; Month 3; Month 4; Month 5; Month 6; Month 7; Month 8; Month 9; Month 10; Month 13; Month 16; Month 19; Month 22; Month 24
  Longitudinal evolution of the score
MADRS (Montgomery-Asberg Depression Rating Scale) | Month -3 ; Month -1; Day -7; Day 15; Month 1; Day 45; Month 2 ; Day 75 ; Month 3; Month 4; Month 5; Month 6; Month 7; Month 8; Month 9; Month 10; Month 13; Month 16; Month 19; Month 22; Month 24
  Longitudinal evolution of the score
BDI (Beck Depression Inventory) | Day -7; Day 15; Month 1; Day 45; Month 2 ; Day 75 ; Month 3; Month 4; Month 5; Month 6; Month 7; Month 8; Month 9; Month 10; Month 13; Month 16; Month 19; Month 22; Month 24
  Longitudinal evolution of the score
CGI (Clinical global impressions) | Month -3 ; Month -1; Day-7; Day15; Month 1; Day 45; Month 2 ; Day 75 ; Month 3; Month 4; Month 5; Month 6; Month 7; Month 8; Month 9; Month 10; Month 13; Month 16; Month 19; Month 22; Month 24
  Longitudinal evolution of the score
LARS (Lille Apathy Rating scale) | Day -7; Month 1; Month 7; Month 13; Month 19; Month 24
  Longitudinal evolution of the score
GAF (Global assessment of functioning) | Month -3 ; Month -1; Day -7; Month 1; Month 7; Month 13; Month 19; Month 24
  Longitudinal evolution of the score
YMRS (Young Mania Rating Scale) | Day -7; Month 1; Month 7; Month 13; Month 19; Month 24
  Longitudinal evolution of the score
MATHYS (Multidimensional Assessment of Thymic States) | Day -7; Month 1; Month 7; Month 13; Month 19; Month 24
  Longitudinal evolution of the score
Response (50 % decrease of the HDRS-17) | Month 24
  During the whole follow up
Remission | M24
  During the whole follow up Remission is defined as an HDRS-17 score < 7

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel Reymann, Study Chair — CIC INSERM 0203 CHU Rennes; Florian Naudet, Study Chair — CIC INSERM 0203 CHU Rennes; Bruno Millet, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (5):
- France (5):
  - APHM, Marseille
  - APHP Pitié Salpetriere, Paris
  - CHS, Poitiers
  - CHS, Rouen
  - CHU, Toulouse